CLINICAL TRIAL: NCT06673472
Title: Comparison of Long-term Outcomes Between Upfront Surgery and Neoadjuvant Therapy Followed by Surgery in Patients with Node-Negative Gastric Cancer: a Propensity Score Matched International Multicenter Study
Brief Title: Comparison of Long-term Outcomes Between Upfront Surgery and Neoadjuvant Therapy Followed by Surgery in Patients with Node-Negative Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Chang-Ming Huang, Prof. (Other)
Responsible Party: Sponsor-Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: 2024KY217
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-09

CONDITIONS: Lymph Node-negative; Gastric Cancer
Keywords: Gastric cancer; Neoadjuvant therapy; Long-term outcomes; Lymph node-negative; SEER database
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients with lymph node-negative gastric cancer, the prognosis of patients who underwent neoadjuvant therapy was poor than that of those who had upfront surgery.

DETAILED DESCRIPTION:
We retrospectively analyzed the clinicopathological data of patients who underwent curative surgery for gastric cancer and were pathologically confirmed to have node-negative metastases between January 2010 and June 2021 at 8 institutions in China. Data from the Surveillance, Epidemiology, and End Results (SEER) database (2004-2020) were used as the validation cohort. The patients were divided into two groups based on whether they received neoadjuvant therapy before surgery: the upfront surgery (UFS) group and the neoadjuvant therapy followed by surgery (NATS) group. A 1:1 propensity score matching analysis was employed to reduce the potential selection bias between the two groups.

ELIGIBILITY:
Inclusion Criteria:

(1) preoperative clinical staging of cT2-4NxM0; (2) primary gastric adenocarcinoma confirmed via pathology; (3) no distant metastasis to the liver, lungs, or abdominal cavity as confirmed through preoperative chest X-ray or chest CT, abdominal ultrasound, and abdominal CT; (4) underwent radical gastrectomy (R0) and D2 lymphadenectomy; (5) postoperative pathology confirmed no lymph node metastasis (i.e., lymph node-negative); and (6) follow-up for at least 3 years.

Exclusion Criteria:

(1) considered early-stage gastric cancer before surgery; (2) distant metastasis detected preoperatively or intraoperatively; (3) failure to achieve R0 resection and D2 lymphadenectomy during surgery; (4) concurrent diagnosis of other malignancies; (5) remnant gastric cancer; (6) death within 30 days postoperatively; and (7) incomplete baseline data or follow-up records.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively analyzed the clinicopathological data of patients who underwent curative surgery for gastric cancer and were pathologically confirmed to have node-negative metastases between January 2010 and June 2021 at 8 institutions in China. Data from the Surveillance, Epidemiology, and End Results (SEER) database (2004-2020) were used as the validation cohort. The patients were divided into two groups based on whether they received neoadjuvant therapy before surgery: the upfront surgery (UFS) group and the neoadjuvant therapy followed by surgery (NATS) group. A 1:1 propensity score matching analysis was employed to reduce the potential selection bias between the two groups.
Sampling Method: Non-Probability Sample
Enrollment: 1081 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
survival | Within 3 years after surgery
  3-year overall survival , disease-specific survival，and disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Chang-ming, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No